CLINICAL TRIAL: NCT06682286
Title: Breathing Route in COPD and OHS Patients on Long-term Home Non-invasive Ventilation: An Experimental Study
Brief Title: Assessment of Breathing Pattern During NIV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: U1111-1308-1838
Record Dates: First submitted 2024-11-05; First posted 2024-11-12 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease); Obesity Hypoventilation Syndrome (OHS)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Obesity Hypoventilation Syndrome

STUDY DESIGN:
Intervention Model Description: Crossover study where the breathing route of each participant will be assessed off- and on NIV. Additionally, the breathing route of each participant on NIV will be investigated during sleep and in awake state.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Breathing route assessment: Awake and off pressure support (No Intervention): Breathing route will be recorded in awake participants without the use of NIV for approximately 30 min.
- Breathing route assessment: Awake and on pressure support (Experimental): Awake participants will be placed on their prescribed pressure support settings and will use two different non-invasive ventilation (NIV) masks, each for about 30 minutes.
  Interventions: Other: NIV mask A; Other: NIV mask B
- Breathing route assessment: Asleep and on pressure support (Experimental): Participants will be placed on their prescribed pressure support settings and will go to sleep. After 60 minutes, they will be awakened to change their mask. They will use two different non-invasive ventilation (NIV) masks, each for a minimum of 60 minutes
  Interventions: Other: NIV mask A; Other: NIV mask B

INTERVENTIONS:
Other: NIV mask A — Bridge free face mask
  Arms: Breathing route assessment: Asleep and on pressure support; Breathing route assessment: Awake and on pressure support
Other: NIV mask B — Full face mask
  Arms: Breathing route assessment: Asleep and on pressure support; Breathing route assessment: Awake and on pressure support

SUMMARY:
COPD and OHS are respiratory conditions that disrupt normal breathing. Positive airway pressure, specifically Non-Invasive Ventilation (NIV), has been shown to improve breathing and reduce symptoms in patients with these conditions. Regular use of NIV can lead to better symptom management, improved quality of life, and reduced use of healthcare resources. The type of mask used for breathing support can greatly affect a patient's comfort and willingness to use it. For conditions like Obstructive Sleep Apnea (OSA), which is a physical blockage of the airway caused by the relaxation of the muscles of the throat, nasal masks are often used because they are comfortable and work well. But for breathing support in the hospital, full face masks are typically used because patients are having significant trouble breathing and tend to breathe through their mouth.

However, it's important to note that we don't yet fully understand the best way to provide breathing support for long-term NIV users, like COPD and OHS patients. The understanding of breathing route is currently only established for OSA. However, conditions like COPD affect the lungs and the overall system used for breathing, which is different from the throat blockage seen in OSA. So, the assumptions we make based on conditions like OSA may not apply to these other conditions. More research is needed to understand this better.

DETAILED DESCRIPTION:
* Participants undergo PSG, lying on their backs while their breathing route is recorded for about 30 minutes.
* The participants are then put on their prescribed airway pressure support with the first randomized mask, and their breathing is recorded again for 30 minutes.
* The mask is switched to the second mask, and the same procedure is repeated.

Participants are then moved to the sleep laboratory for the night where they are provided with beds.

* They continue NIV therapy with the last mask used during the awake test.
* After at least 60 minutes of recording, participants are awakened to switch back to the first mask. They are then allowed to sleep uninterrupted for the rest of the night.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Prescribed nocturnal NIV for COPD or OHS
* Able to complete an overnight sleep study
* Comfortable to sleep on a standard double bed
* Capacity to complete informed consent

Exclusion Criteria:

* Uncontrolled sleep apnea (Apnea-hypopnea index (AHI) over 15 events/hour off personal NIV device data)
* Prescribed IPAP above 25 cmH2O
* Self-reported pregnancy
* Allergic to adhesive of the sensors
* Self-reported cold/flu symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-24 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Breathing route while on and off pressure support (awake) | 4 hours
  Percent of time nose and mouth breathing in COPD and/or OHS patients while on and off pressure support.
Breathing route while on pressure support (asleep) | 8 hours
  Percent of time nose and mouth breathing in COPD and/or OHS patients while on pressure support during sleep.
Mask type influence on breathing route (asleep and awake) | 12 hours
  Percent of time nose and mouth breathing in COPD and/or OHS patients depending on the NIV mask type

CONTACTS AND LOCATIONS:
Overall Officials: William Good, Medical degree, Principal Investigator — Middlemore Hospital, New Zealand
Locations (1):
- Fisher and Paykel Healthcare Sleep Laboratory, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No